CLINICAL TRIAL: NCT00437177
Title: Relationship Between D2 Receptors SPECT and the Apomorphine Test in Patients With OH Dependence: Predictive Value for Relapse
Brief Title: Relationship Between D2 Receptors SPECT and the Apomorphine Test in Patients With OH Dependence (ALC-DRD2-APO)
Acronym: ALC-DRD2-APO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: m, Servei de Psiquiatria. Hospital Universitari Vall d'Hebron
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OH SPECT APO; EudraCT: 2004-001893-24
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Alcoholism
Keywords: alcoholism; apomorphine; iodobenzamide; imaging; spect; relapse
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Apomorphine; Iodine-123

INTERVENTIONS:
Drug: apomorphine — Apomorphine 0.05 mg/kg subcutaneously at hospital admission and at discharge. Abstinent participants at 3 months will receive a third dose.
Drug: [(123)I] iodobenzamide — [(123)I] iodobenzamide 185 MBq I.V., at discharge.

SUMMARY:
OH dependence is associated with DA receptor changes. Both, the apomorphine test and the D2Rec SPECt are usefull for monitoring DA receptor status. We aimed at studying whether DA receptor hypofunction, assessed by means of the apomorphine test and the D2Rec SPECT, is a marker of relapse in detoxified OH dependents patients.

ELIGIBILITY:
Inclusion Criteria:

* alcohol dependence
* alcohol dependence length at least 8 years.
* male
* age 25 - 60 years

Exclusion Criteria:

* other drug dependence (except nicotine dependence)
* another major axis I psychiatric diagnosis
* comorbid neurological disorder
* comorbid cardiovascular disorder
* comorbid metabolic disorder
* brain injury
* apomorphine allergy
* iode allergy
* diazepam allergy

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To detertmine the agreement rate of the dopaminergic sensibility assessed by two different techiniques: the apomorphine test and and IBZM SPECT. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Casas, Prof, Principal Investigator — Psychiatry Service, Hospital Universitari Vall d'Hebron
Locations (1):
- Psychiatry Service, Hospital Universitari Vall d'Hebron, Barcelona, Catalonia, Spain